CLINICAL TRIAL: NCT05574855
Title: Echocardiographic and Ultrasound Evaluation of Haemodynamic Parameters in Hypoxic Neonates Treated With Hypothermia.
Brief Title: Evaluation of Haemodynamic in Neonates Treated With Hypothermia"
Status: Completed | Type: Observational
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Renata Bokiniec, MD, Clinical Professor, Head of Department of Neonatology, Princess Anna Mazowiecka Hospital, Warsaw, Poland
Other Study IDs: 0048225966136
Record Dates: First submitted 2022-09-30; First posted 2022-10-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hypothermia Neonatal; Haemodynamic Instability; Perinatal Asphyxia
Keywords: Echocardiography; Neonate; Perinatal asphyxia; Therapeutic hypothermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I study (SG): Neonates with gestational age ≥35, who experienced an episode of perinatal ischaemia and who were qualified for hypothermia treatment according to the Standards of Medical care of Neonates in Poland will be enrolled to the study group (SG) ( n=58)
  Initial echocardiography and cerebral and abdominal ultrasonography were performed at two key time points:
  No echo were performed on passive TH.
  1. Since qualification for TH takes place up to 6 hours of life (HOL), the first examination in the SG took place between 6 and 54HOL after reaching a body temperature of 33.5°C (SG1).
  2. The second examination (SG2) was performed after the TH procedure was completed and after the RW, when the body temperature reached 36.6°C, i.e., after 90HOL, but no later than 7DOL.
- Group II controls (CG): Healthy term neonates who underwent ECHO due to difficult adaptation or maternal gestational diabetes were enrolled in CG1 (n=14), and those who underwent ECHO after ductus arteriosus closure or with only a trace, hemodynamically insignificant ductus, were enrolled in CG2(n=44).
  Initial echocardiography and cerebral and abdominal ultrasonography were performed at two key time points:
  1. Health term neonates who were enrolled to the CG1 underwent ECHO at the 1/2DOL ( n=14)
  2. Those who were enrolled to the CG2 underwent ECHO between 3 and 7 DOL.(n=44)

SUMMARY:
Perinatal hypoxia in the form of hypoxic-ischaemic encephalopathy (HIE) is a frequent cause of cerebral impairment in neonates. HIE occurs in 3 to 5 of 1000 neonates in developed countries and is significantly higher in developing countries at 25 of 1000 neonates. Despite developments in medicine, increasing understanding of HIE pathophysiology and progress in neonatal intensive care as well as treatment of moderate or severe perinatal asphyxia, HIE continues to be associated with significant mortality and late neurological sequelae.

Episodes of ischaemia-hypoxia in the perinatal period as well as the changes in the redistribution of blood may lead to decreased perfusion and ischaemia of the cardiac muscle. Additionally, there is a negative impact from the reduced contractility of the cardiac muscle secondary to acidosis and hypoxia. Therapeutic hypothermia (TH) improves the late effects in moderate and severe cases of hypoxia-ischaemia encephalopathy (HIE). The direct impact of TH on the cardiovascular system includes moderate bradycardia, increased pulmonary vascular resistance (PVR), inferior filling of the left ventricle (LV) and LV stroke volume. The above-mentioned consequences of TH and episodes of HI in the perinatal period are therefore exacerbation of respiratory and circulatory failure. The impact of the warming phase on the cardiovascular system is not well researched and currently few data has been published on this topic. Physiologically, warming increases heart rate, improves cardiac output and increases systemic pressure. The effect of TH and the warming phase on the cardiovascular values has a decisive impact on the metabolism of drugs, including vasopressors / inotropics, which in turn affects the choice of medication and fluid therapy

DETAILED DESCRIPTION:
Impact of hypoxia on the cardiovascular system Transitory hypoxia of the myocardium (and its resultant dysfunction), which may, but not necessarily, present clinically, occurs in two thirds of neonates born with perinatal asphyxia. There is no doubt that that this is one of the more frequent cause of circulatory insufficiency. Both an episode of ischaemic hypoxia in the perinatal period and the changes in the distribution of blood may lead to diminished perfusion of the cardiac muscle. An additional but no less important impact on cardiac function is the immaturity of the neonatal myocardium and its reduced contractility secondary to acidosis and hypoxia. Ischaemia and acidosis lead to imbalance in favour of production of endothelin 1, which leads to reduced production of nitric oxide and vasoconstriction of pulmonary vessels and therefore greater pulmonary vascular resistance (PVR) which has a detrimental effect on the already impaired right ventricular (RV) function. The weak RV function and increase PVR impair filling and function of the left ventricle (LV) and thus, they can affect systemic and cerebral blood flow.

The impact of therapeutic hypothermia on the cardiovascular system

TH improves the distant results in cases of moderate and severe HIE and is currently the standard of care for neonates born at or near term (> 35 weeks of gestation). The direct effect of TH on the cardiovascular system includes the following:

* Moderate bradycardia resulting from the decreased effect of the parasympathetic system on cardiac function. Indeed, sinus bradycardia leads to reduced stroke volume and decreased requirement for energy by the myocardium. In turn, administration of inotropes increase metabolic requirements.
* Additionally, TH leads to increased PVR, potentially resulting in a clinical picture of persistent pulmonary hypertension in the neonate (PPHN) or its exacerbation in cases of pre-existing raised PVR. In animal studies, TH was associated with increased PVR, while an increased risk of PPHN with TH was not found in RCTs.
* The resulting RV dysfunction and reduced stroke capacity of the RV leads to reduced pulmonary venous return and therefore inferior filling and stroke volume of the LV. A consequence of the effects of TH mentioned above and of an episode of HI in the perinatal period is therefore exacerbation of respiratory and circulatory failure.

Impact of the warming process on the cardiovascular system following administration of hypothermia

The impact of the warming phase on the cardiovascular system has not been well documented and currently very little data was published on this topic. Physiologically warming accelerates the heartbeat and improves stroke volume, although the mean blood pressure may fall or remain unchanged as a result of lowering of the diastolic component, which in turn affects metabolism and drug clearance, including clearance of cardiovascular medications. The warming phase, following conclusion of hypothermic treatment, affects the selection of further medicinal therapy in terms of vasopressors, inotropes and of fluid therapy. Furthermore, studies have shown that neonates are more at risk of convulsive episodes during the warming phase. In a study of 160 neonates, 9% experienced intra- or periventricular haemorrhage. Neonates require more precise observation in terms of haemodynamic instability during the warming phase.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates with gestation age ≥35, whith episode of PA and who were qualified for TH according to the Standards of Medical care of Neonates in Poland (10) was enrolled to the SG
2. Healthy, neonates with gastation >37 0/7 < 41 6/7, who underwent ECHO for reasons such as difficult adaptation, gestational diabetes of the mother etc. was enrolled to the CG.

Exclusion Criteria:

1. Congenital cardiac abnormalities
2. Genetic abnormalities
3. Absence of parental or guardian consent for participation in the study
4. SGA <10 centiles

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a multicentre, prospective, case-control, observational study. The number of subjects under observation will be 113 neonates. The enrolment, intervention and assessment schedule is presented in tabel.
  Initial echocardiography and cerebral and abdominal ultrasonography will be conducted according to physician recommendation by two neonatologist.
  The study procedure will be explained to patient's guardians who will also receive an information leaflet. Guardians will then be asked to provide two copies of informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Assessment of the influence of Therapeutic hypothermia (TH) on systolic-diastolic functions of the left ventricles in comparison with the control group using the Pulse Doppler | until 7 day after birth
  LV systolic and diastolic function on cardiac echocardiography will be assessed using the Pulse Doppler
Assessment of the influence of Therapeutic hypothermia (TH) on systolic-diastolic functions of the right ventricles in comparison with the control group using the Pulse Doppler | until 7 day after birth
  RV systolic and diastolic function on cardiac echocardiography will be assessed using the Pulse Doppler
Assessment of the influence of Therapeutic hypothermia (TH) on systolic-diastolic functions of the left ventricles in comparison with the control group using the M-mode. | until 7 day after birth
  LV systolic and diastolic function on cardiac echocardiography will be assessed using the M-mode.
Assessment of the influence of Therapeutic hypothermia (TH) on systolic-diastolic functions of the right ventricles in comparison with the control group using the M-mode. | until 7 day after birth
  RV systolic and diastolic function on cardiac echocardiography will be assessed using the M-mode.
Assessment of the effect of the warming phase on the systolic-diastolic functions of the left ventricles in comparison with the control group using the Tissue Doppler | until 7 day after birth
  LV systolic and diastolic function on cardiac echocardiography will be assessed using the Tissue Doppler
Assessment of the effect of the warming phase on the systolic-diastolic functions of the right ventricles in comparison with the control group using the Tissue Doppler | until 7 day after birth
  RV systolic and diastolic function on cardiac echocardiography will be assessed using the Tissue Doppler

SECONDARY OUTCOMES:
Assessment of the influence of TH on the cerebral circulation in comparison with the control group in arterior cerebral artery | until 7 day after birth
  Controls cerebral circulation in neonates by Doppler evaluation of blood flow in anterior cerebral artery(ACA),
Assessment of the influence of TH on the cerebral circulation in comparison with the control group in middle cerebral artery | until 7 day after birth
  Assessment of cerebral circulation in neonates and controls by Doppler evaluation of blood flow in middle cerebral artery (MCA),
Assessment of the influence of TH on the cerebral circulation in comparison with the control group in the superior vena cava | until 7 day after birth
  Assessment of cerebral circulation in neonates and controls by Doppler evaluation of blood flow in the superior vena cava - SVC (CO)
Assessment of the influence of TH on the visceral circulation in comparison with the control group | until 7 day after birth
  Assessment of visceral circulation in neonates and controls by Doppler blood flow evaluation in mesenteric artery (SMA).
Assessment of the influence of TH on the renal circulation in comparison with the control group | until 7 day after birth
  Assessment of renal circulation in neonates and controls by Doppler blood flow evaluation in right renal artery (RRA).
Assessment of the effect of the warming phase on the cerebral circulation in comparison with the control group in arterior cerebral artery | until 7 day after birth
  Assessment of cerebral circulation in neonates and controls by Doppler evaluation of blood flow in anterior cerebral artery (ACA)
Assessment of the effect of the warming phase on the cerebral circulation in comparison with the control group in middle cerebral artery | until 7 day after birth
  Assessment of cerebral circulation in neonates and controls by Doppler evaluation of blood flow in middle cerebral artery (MCA)
Assessment of the effect of the warming phase on the cerebral circulation in comparison with the control group in the superior vena cava | until 7 day after birth
  Assessment of cerebral circulation in neonates and controls by Doppler evaluation of blood flow in the superior vena cava - SVC (CO)
Assessment of the effect of the warming phase on the visceral circulation in comparison with the control group | until 7 day after birth
  Assessment of visceral circulation in neonates and controls by Doppler blood flow evaluation in mesenteric artery (SMA.)
Assessment of the effect of the warming phase on the renal circulation in comparison with the control group | until 7 day after birth
  Assessment of renal circulation in neonates and controls by Doppler blood flow evaluation in right renal artery (RRA.)

CONTACTS AND LOCATIONS:
Locations (4):
- Poland (4):
  - Department of Neonatology and Neonatal Intensive Care Warsaw Medical University, Warsaw
  - Princess Anna Mazowiecka Hospital, Warsaw
  - Centrum Medyczne "ŻELAZNA", Warsaw
  - Lazarski University Faculty of Medicine, Warsaw

REFERENCES:
- [Background] Yoon JH, Lee EJ, Yum SK, Moon CJ, Youn YA, Kwun YJ, Lee JY, Sung IK. Impacts of therapeutic hypothermia on cardiovascular hemodynamics in newborns with hypoxic-ischemic encephalopathy: a case control study using echocardiography. J Matern Fetal Neonatal Med. 2018 Aug;31(16):2175-2182. doi: 10.1080/14767058.2017.1338256. Epub 2017 Jul 7. PMID 28573895
- [Background] Wu TW, Tamrazi B, Soleymani S, Seri I, Noori S. Hemodynamic Changes During Rewarming Phase of Whole-Body Hypothermia Therapy in Neonates with Hypoxic-Ischemic Encephalopathy. J Pediatr. 2018 Jun;197:68-74.e2. doi: 10.1016/j.jpeds.2018.01.067. Epub 2018 Mar 20. PMID 29571928
- [Background] Sehgal A, Linduska N, Huynh C. Cardiac adaptation in asphyxiated infants treated with therapeutic hypothermia. J Neonatal Perinatal Med. 2019;12(2):117-125. doi: 10.3233/NPM-1853. PMID 30814366
- [Background] Bhagat I, Sarkar S. Multiple Organ Dysfunction During Therapeutic Cooling of Asphyxiated Infants. Neoreviews. 2019 Nov;20(11):e653-e660. doi: 10.1542/neo.20-11-e653. PMID 31676739
- [Derived] Brunets N, Brunets V, Bokiniec R. Echocardiographic and ultrasound evaluation of haemodynamic parameters in hypoxic neonates treated with hypothermia: Study protocol. Front Pediatr. 2023 Apr 18;11:1122738. doi: 10.3389/fped.2023.1122738. eCollection 2023. PMID 37144150